CLINICAL TRIAL: NCT06072716
Title: The Anti-fungal Effect of Miconazol and Miconazol-Loaded Chitosan Nanoparticles in Diabetic Patients With Oral Candidiasis-Randomized Control Clinical Trial and Microbiological Analysis
Brief Title: The Anti-fungal Effect of Miconazol Versus Miconazol-Loaded Chitosan Nanoparticles
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yasmine gamil (Other)
Responsible Party: Sponsor-Investigator, Yasmine gamil, Lecturer of oral medicine and diagnosis, MTI University
Organization: MTI University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mti University
Record Dates: First submitted 2023-09-21; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Oral Thrush
Keywords: diabetic patients or oral candidiasis or oral thrush
MeSH Terms: conditions — Candidiasis; Candidiasis, Oral | interventions — Chitosan

STUDY DESIGN:
Intervention Model Description: 1:1 parallel arms
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional (Experimental): chitosan loaded with miconazole nanoparticles gel
  Interventions: Drug: Chitosan
- control (Experimental): miconazole gel
  Interventions: Drug: Chitosan

INTERVENTIONS:
Drug: Chitosan — chitosan loaded with miconazole nanoparticles gel
  Other Names: miconaz oral gel

SUMMARY:
Objective: this study aimed to evaluate the therapeutic effects of topical application of miconazole and miconazole-loaded chitosan nanoparticles in treatment diabetic patients with oral candidiasis.

DETAILED DESCRIPTION:
Abstract:

Objective: this study aimed to evaluate the therapeutic effects of topical application of miconazole and miconazole-loaded chitosan nanoparticles in treatment diabetic patients with oral candidiasis.

Subjective and methods:

In this randomized controlled clinical trial,. A total of 80 diabetic patients presenting with symptomatic oral candidiasis were randomly assigned into two treatment groups: miconazole and miconazole-loaded chitosan nanoparticles. The patients were treated for a duration 28days , and clinical assessments were conducted at baseline, 7, 14, 21 and 28 days.

Microbiological analysis was performed to determine the Candida species and assess their susceptibility to the antifungal agents. Clinical parameters, including signs and symptoms of oral candidiasis, were also evaluated.

.

ELIGIBILITY:
Inclusion Criteria:

1. uncontrolled diabetes patients with oral candidiasis and their uncontrolled diabetes were confirmed by doing glycated hemoglobin test and their range is >7.0%,
2. age ranged from 30-65 years
3. patients were willing to participate in this study

Exclusion Criteria:

1. immunocompromised and patients with systemic diseases that can cause muscle weakness as Parkinson's disease, or others that can limit their cognitive functioning such as dementia
2. pregnant
3. nursing women
4. smokers
5. alcoholic patients were also excluded from the study.
6. should not have a history of use of any drugs that can cause hyposalivation or broad spectrum antibiotics, within the last month.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
clinical assessment of erythematous/psuedomembranous oral candidiasis resolution | 28 days
  by Pain analogue scale

SECONDARY OUTCOMES:
microbiological count of candida | 28 days
  candidal count by taking swap

CONTACTS AND LOCATIONS:
Overall Officials: radwa ELsherif, PHD, Principal Investigator — MUST
Locations (1):
- radwa Elsherif, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gamil Y, Hamed MG, Elsayed M, Essawy A, Medhat S, Zayed SO, Ismail RM. The anti-fungal effect of miconazole and miconazole-loaded chitosan nanoparticles gels in diabetic patients with Oral candidiasis-randomized control clinical trial and microbiological analysis. BMC Oral Health. 2024 Feb 7;24(1):196. doi: 10.1186/s12903-024-03952-0. PMID 38321454